CLINICAL TRIAL: NCT02214082
Title: Feasibility and Safety of Same Day Discharge After Elective Percutaneous Coronary Intervention (PCI) in a Tertiary Care Hospital in Karachi, Pakistan.
Brief Title: Safety of Same Day Discharge After Elective Percutaneous Coronary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indus Hospital and Health Network (Other)
Responsible Party: Principal Investigator, Sajid H. Dhakam, Faculty, Cardiology, Indus Hospital and Health Network
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIH-Cardio-001
Record Dates: First submitted 2014-08-09; First posted 2014-08-12 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Angioplasty; Coronary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Next day discharge (No Intervention): this group will be discharged as is the standard practice at our facility; i.e. the day after the PCI procedure
- Same Day Discharge (Experimental): Patients in this arm will be discharged on the same day as their angioplasty.
  Interventions: Other: Same Day Discharge

INTERVENTIONS:
Other: Same Day Discharge — This group will be discharged home, on the same day after their elective angioplasty
  Arms: Same Day Discharge

SUMMARY:
Study intends to determine if there is any difference in the occurrence of major adverse cardiology events in patients discharged on the same day as their elective cardiac angioplasty or discharged one day after their angioplasty.

Hypothesize that same day discharge is as safe as a day later discharge.

ELIGIBILITY:
Inclusion Criteria: :

* Low risk lesion (according to the ACC classification)
* Normal Pre Catheterization laboratory investigation
* Procedure performed before 3 pm
* procedure performed with ≤ 6 French guiding Catheter
* EF ≥ 35%
* living at a distance of within 15 kilometers from hospital
* caregiver present at home
* elective procedure

Exclusion Criteria:

* Acute PCI
* high risk lesions (according to the ACC classification)
* deranged Pre Catheterization laboratory investigations
* Age >70
* Severe LV dysfunction, CVA
* procedure to be performed with a guiding catheter >6F
* Use of IIb/IIIa inhibitor
* Creatinine clearance of < 50

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mortality | Within 30 days post angioplasty
Number of patients who require a 2nd angioplasty | within 30 days of 1st angioplasty
Number of patients with bleed from the angioplasty site | within 30 days post angioplasty

SECONDARY OUTCOMES:
number of hospital re-admissions | within 30 days of initial angioplasty

CONTACTS AND LOCATIONS:
Overall Officials: Sajid Dhakam, Principal Investigator — Indus Hospital and Health Network
Locations (1):
- The Indus Hospital, Karachi, Sindh, Pakistan